CLINICAL TRIAL: NCT06578182
Title: The Effect of ColcHicine on the Incidence of Knee or Hip Replacements: a Randomized, Double-blind, Multicentre Study in Symptomatic Knee or Hip Osteoarthritis
Brief Title: The Effect of ColcHicine on the Incidence of Knee or Hip Replacements
Acronym: ECHO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); RSMK (Unknown); Tiofarma (Unknown); Dutch Arthritis Foundation Reuma Nederland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMaartenskliniek; 10140262210012 (Other Grant/Funding Number: ZonMW); 2024-511359-16-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-04; First posted 2024-08-29 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Colchicine; Knee replacement; Hip replacement
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Experimental)
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — Colchicine 0.5mg tablets once a day for 3 to 4.5 years
  Arms: Colchicine
Drug: Placebo — Placebo tablets once a day for 3 to 4.5 years
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the effect of treatment with colchicine 0.5mg once daily as compared to placebo in patients with knee or hip osteoarthritis on the incidence of first occurrence of knee or hip replacement. The main question it aims to answer is:

Does colchicine lower the number of knee or hip replacements in participants with osteoarthritis?

Researchers will compare colchicine to a placebo (a look-alike substance that contains no drug) to see if colchicine works to treat osteoarthritis.

Participants will:

* take colchicine every day for 3 tot 4.5 years
* visit the clinic every year for check-up and tests such as blood samples and x-rays
* fill in questionnaires every 3 months

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of knee or hip OA
* 45 ≤ age ≤ 80 (upper age limit is similar to that in the LoDoCo2 trial and takes in consideration the lower number of joint replacements in people older than 80 years)
* documented radiographic changes typical for advanced knee/hip OA (Kellgren & Lawrence score ≥ 2), or at least 2-year history of complaints due to OA in the hip and/or knee

Exclusion Criteria:

* On a waiting list for primary joint replacement surgery of the hip or knee, irrespective of cause
* Any absolute contraindication for knee or hip replacement in the future
* More than one previous hip or knee replacements
* Other known medical disease that may affect joints
* Known generalized pain syndromes such as fibromyalgia
* Renal impairment as evidenced by serum creatinine >150µmol/l or estimated glomerular filtration rate (eGFR) <50mL/min/1.73m2
* Liver function impairment as evidenced by serum alanine transferase (ALAT) > 3 ULN (upper limit of normal)
* Blood dyscrasia
* High frailty (clinical frailty scale ≥ 7) or predicted life expectancy < 5 years
* Peripheral neuritis, myositis or marked myo-sensitivity to statins
* Current use of colchicine for another indication
* Intolerance to colchicine
* use of macrolide antibiotics (i.e. clarithromycin, erythromycin, azithromycin), antimycotics (i.e. ketoconazole, itraconazole and voriconazole), protease inhibitors & anti-retroviral drugs (i.e. ritonavir, lopinavir, tipranavir, atazanavir, darunavir, indinavir, saquinavir, and cobicistat), anti-arrhythmic drugs (i.e. verapamil, diltiazem), or immunosuppressant (i.e. cyclosporine)
* Current enrollment in another trial
* Incapacitated patients
* Pregnant or breastfeeding female
* Fertile female participants not taking sufficient anti-conception
* Male participants unwilling to use effective contraception during the study to prevent pregnancy

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1410 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Time to first knee or hip replacement | From randomization until the date of first documented knee or hip replacement, date of death, date of lost to follow-up, or study end-date, whichever comes first, assessed up to 4.5 years

SECONDARY OUTCOMES:
Course of pain as assessed by NRS (numeric rating scale) | From randomization until the date of first documented knee or hip replacement, date of death, date of lost to follow-up, or study end-date, whichever comes first, assessed up to 4.5 years
  The 11-point NRS ranges from '0' ("no pain") to '10' ("worst pain imaginable")
Course of pain as assessed by WOMAC (Western Ontario and McMaster Universities Arthritis Index) | From randomization until the date of first documented knee or hip replacement, date of death, date of lost to follow-up, or study end-date, whichever comes first, assessed up to 4.5 years
  5 items are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). Higher scores indicate more pain
Course of physical function as assessed by WOMAC (Western Ontario and McMaster Universities Arthritis Index) | From randomization until the date of first documented knee or hip replacement, date of death, date of lost to follow-up, or study end-date, whichever comes first, assessed up to 4.5 years
  17 items are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). Higher scores indicate more functional limitations
Course of joint space narrowing on X-ray | From baseline until the date of first documented knee or hip replacement or study end, whichever comes first, assessed up to 4.5 years
Course of low-grade inflammation as assessed by hs-CRP | At enrolment, at baseline, 1 year thereafter, and at study completion (approximately 4.5 years)
Course of quality of life as assessed by EQ-5D-5L (European Quality of Life 5 Dimensions) | From randomization until the date of first documented knee or hip replacement, date of death, date of lost to follow-up, or study end-date, whichever comes first, assessed up to 4.5 years
  The EQ-5D-5L comprises 5 dimensions with each dimension having 5 response levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4), unable to/extreme problems (5). EQ-5D-5L health states can be represented by a single summary number (index value) (range -0.624 to 1.000). Higher scores equals better quality of life
Number of participants with clinical or radiological onset of OA in new joint group other than present at baseline over the trial period | From randomization until the date of first documented knee or hip replacement, date of death, date of lost to follow-up, or study end-date, whichever comes first, assessed up to 4.5 years
Time to clinical or radiological onset of OA in new joint group other than present at baseline over the trial period | From randomization until the date of first documented knee or hip replacement, date of death, date of lost to follow-up, or study end-date, whichever comes first, assessed up to 4.5 years
Number of participants using pain medication during the study registered per drug type (e.g. paracetamol, NSAIDs, opioids) | From randomization until the date of first documented knee or hip replacement, date of death, date of lost to follow-up, or study end-date, whichever comes first, assessed up to 4.5 years
Onset of new cardiovascular events, defined as myocardial infarction, peripheral artery disease, ischemia-driven coronary revascularization, ischemic stroke, or cardiovascular death | From randomization until the date of first documented knee or hip replacement, date of death, date of lost to follow-up, or study end-date, whichever comes first, assessed up to 4.5 years
Direct and indirect costs related to treatment and disease burden due osteoarthritis | From randomization until the date of first documented knee or hip replacement, date of death, date of lost to follow-up, or study end-date, whichever comes first, assessed up to 4.5 years

OTHER OUTCOMES:
The number of (serious) adverse events | From randomization until the date of first documented knee or hip replacement, date of death, date of lost to follow-up, or study end-date, whichever comes first, assessed up to 4.5 years
  Adverse events are defined as any untoward medical occurrence in a subject to whom a medicinal product is administered, and which does not necessarily have a causal relationship with this treatment.
  Serious adverse event is any untoward medical occurrence in a patient or trial subject that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect
The number of withdrawals due to (serious) adverse events | From randomization until the date of first documented knee or hip replacement, date of death, date of lost to follow-up, or study end-date, whichever comes first, assessed up to 4.5 years
  Adverse events are defined as any untoward medical occurrence in a subject to whom a medicinal product is administered, and which does not necessarily have a causal relationship with this treatment. Serious adverse event is any untoward medical occurrence in a patient or trial subject that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect
Changes in laboratory data (i.e. serum creatinine, estimated glomerular filtration rate, and alanine transferase) | At enrolment, at baseline, 1 year thereafter, and at study completion (approximately 4.5 years)

CONTACTS AND LOCATIONS:
Locations (1):
- Sint Maartenskliniek, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heijman MWJ, van den Ende CHM, Cornel JH, Smolders JMH, Schers HJ, Kievit W, Koeter S, van den Bemt BJF, Popa CD. Design of a randomised, placebo-controlled, double-blind multicentre study assessing the effect of colchicine on the incidence of knee or hip replacements in symptomatic knee or hip osteoarthritis: the ECHO trial. BMJ Open. 2025 Apr 14;15(4):e098096. doi: 10.1136/bmjopen-2024-098096. PMID 40228852